CLINICAL TRIAL: NCT05782088
Title: Single Versus Repeated Piezocision-assisted Orthodontic Tooth Movement: a Randomized Controlled Clinical Trial
Brief Title: Single Versus Repeated Piezocision-assisted Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Orthodontic Tooth Movement; Canine Retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Piezocision (Experimental)
  Interventions: Procedure: Single Piezocision
- Repeated Piezocision (Experimental)
  Interventions: Procedure: Repeated Piezocision

INTERVENTIONS:
Procedure: Single Piezocision — Piezocision will be performed only once before the onset of canine retraction (T0) on one side of the maxillary arch that will be randomly chosen.
  Arms: Single Piezocision
Procedure: Repeated Piezocision — Piezocision will be repeated three times, on a monthly basis (T0, T1, and T2), over the 12-week study period.
  Arms: Repeated Piezocision

SUMMARY:
The primary aim of the study is to evaluate the effect of single and repeated piezocisions on the rate of orthodontic tooth movement. Secondary aims are to evaluate the effect of both protocols on molar anchorage loss, as well as on canine root resorption.

ELIGIBILITY:
Inclusion Criteria:

* Malocclusion that requires at least the extraction of maxillary first premolars, such as Class I bimaxillary protrusion, and Class II division 1 cases.
* Normal shape and structure of the maxillary canines, with no history of root canal treatment

Exclusion Criteria:

* Patients who underwent previous orthodontic treatment.
* Patients currently receiving drug therapy that may affect orthodontic tooth movement, e.g. hormonal therapy and corticosteroids.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Measurement of canine retraction | 12 weeks
  Several landmarks will be identified on the dental arch, including the mid-palatal raphe, the most medial points on the third right and left rugae, and the cusp tips of the right and left maxillary canines. Perpendicular lines will be drawn from the medial points of the right and left third rugae, and the cusp tips of the right and left maxillary canines to the mid-palatal raphe. The antero-posterior measurements will be carried out between the canine lines and the third rugae lines bilaterally, to assess the rate of canine retraction.
Measurement of molar anchorage loss | 12 weeks
  Perpendicular lines will be drawn from the central fossae of both maxillary right and left first molars to the mid-palatal raphe. Consequently, molar anchorage loss will be calculated by measuring the distance between those lines, and the lines representing the third rugae as previously mentioned.
Measurement of canine root resorption | 12 weeks
  Root resorption of the maxillary canines will be evaluated and measured by comparing pre-retraction and post-retraction CBCT scans.
Bone Microstructure (Fractal Dimension) | 12 weeks
  Using the collected CBCT scans, the region of interest will be selected within the maxillary alveolar process, and the fractal dimension analysis will be performed using a special software for the maxillary canines in the experimental and control groups.
Alveolar bone density | 12 weeks
  From the acquired pre- and post-retraction CBCTs, bone density will be measured form a coronal cross-section of the maxillary arch around each canine in the experimental and control groups.
Alveolar bone thickness | 12 weeks
  The buccal bone thickness will also be measured at three points from the buccal bone to the root, at the coronal, mid-root, and apical level for each maxillary canine
Alveolar bone volume | 12 weeks
  From the pre- and post-retraction CBCTs (at T0 and T1), bone volume in areas of the maxillary alveolar process surrounding the canines will be measured using a special software.
Maxillary canine tipping | 12 weeks
  Tipping of the maxillary canine during retraction was evaluated by drawing vertical lines on the palatal surfaces of the lateral incisor and the canine that extend from the middle of the incisal edge of the lateral incisor and the cusp tip of the maxillary canine to the middle of the cervical line of each, thereby dividing each of them into equal halves. The distance between the lateral incisor and the canine was assessed at two points on their clinical crowns: incisal, and cervical, enabling the detection of crown tipping of the canine during retraction if there was a difference in the measurements between the both the assessed levels.

CONTACTS AND LOCATIONS:
Overall Officials: Farah Y Eid, PhD, Principal Investigator — Alexandria University; Ahmed R El-Kalza, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Eid FY, El-Kalza AR. The effect of single versus multiple piezocisions on the rate of canine retraction: a randomized controlled trial. BMC Oral Health. 2024 Aug 30;24(1):1024. doi: 10.1186/s12903-024-04716-6. PMID 39215274